CLINICAL TRIAL: NCT00763659
Title: Long Term Effects of Lutein/Zeaxanthin and Omega-3- Supplementation on Optical Density of AMD Patients (LUTEGA)
Acronym: LUTEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Jens Dawczynski, Prof. Dr. med. jens Dawczynski, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2032-06/07
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Age Related Maculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 20mg Lutein, 2mg Zeaxanthin, 510 mg Omega-3-FA; daily supplementation about one year
  Interventions: Dietary Supplement: Lutein/ Zeaxanthin + Omega-3-FA
- 2 (Active Comparator): 10mg Lutein, 1mg Zeaxanthin, 255 mg Omega-3-FA; daily supplementation about one year
  Interventions: Dietary Supplement: Lutein/ Zeaxanthin + Omega-3-FA
- 3 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lutein/ Zeaxanthin + Omega-3-FA — 20mg Lutein, 2mg Zeaxanthin, 510 mg Omega-3-FA; daily supplementation about one year
  Arms: 1
Dietary Supplement: Lutein/ Zeaxanthin + Omega-3-FA — 10mg Lutein, 1mg Zeaxanthin, 255 mg Omega-3-FA; daily supplementation about one year
  Arms: 2
Dietary Supplement: Placebo — 0 mg Lutein, Zeaxanthin, Omega-3-FA
  Arms: 3

SUMMARY:
The primary objective of LUTEGA is it to determine the long term effect (about 1 year) of the supplementation with a fixed combination of lutein/zeaxanthin and omega-3- fatty acids on the optical density (OD) of macular pigment in patients with non- exudative age related maculopathy.

Furthermore, it is to be examined whether changes of the optical density are different dosages dependent. Possible changes of lipofuscin content and effect on drusen in AMD patients are studied. The measurement of optical density of macular pigment uses the 1- wavelength reflection method recording reflection images at 460 nm by a fundus camera. The patients are investigated at baseline and are followed up over one year in four more visits. In addition to the OD- measurement each examination includes standardized visual acuity test (ETDRS), amsler- grid, slit lamp biomicroscopy, fundus photography (color and autofluorescence) and a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* All non- exudative forms of age related maculopathy

Exclusion Criteria:

* Exudative age related maculopathy

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Optical density of macular pigment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Strobel, MD, Study Director — University Hospital, Jena; Jens Dawczynski, MD, Principal Investigator — University Hospital, Jena
Locations (1):
- Department of Ophthalmology, University Hospital, Jena, Germany

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300
- [Derived] Dawczynski J, Jentsch S, Schweitzer D, Hammer M, Lang GE, Strobel J. Long term effects of lutein, zeaxanthin and omega-3-LCPUFAs supplementation on optical density of macular pigment in AMD patients: the LUTEGA study. Graefes Arch Clin Exp Ophthalmol. 2013 Dec;251(12):2711-23. doi: 10.1007/s00417-013-2376-6. Epub 2013 May 22. PMID 23695657
- [Derived] Arnold C, Winter L, Frohlich K, Jentsch S, Dawczynski J, Jahreis G, Bohm V. Macular xanthophylls and omega-3 long-chain polyunsaturated fatty acids in age-related macular degeneration: a randomized trial. JAMA Ophthalmol. 2013 May;131(5):564-72. doi: 10.1001/jamaophthalmol.2013.2851. PMID 23519529